CLINICAL TRIAL: NCT06097104
Title: The Incidence, Risk Factors and Outcomes of Electrolytes Disturbances in Critically Ill Egyptian Patients: A Single-Centre Prospective Cohort Study
Brief Title: Electrolytes Disturbances in Critically Ill Egyptian Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: FMASU MD195/2023
Record Dates: First submitted 2023-10-05; First posted 2023-10-24 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-04

CONDITIONS: Electrolyte Imbalance
Keywords: Electrolytes; Egyptian

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: electrolytes - serum blood samples — CBC - Kidney function tests - liver function tests - ABG - levels of serum sodium, potassium, magnesium, phosphorus, ionized calcium and chloride", with maximum 5 mm blood sampling per day

SUMMARY:
All selected individuals will be subjected to the following:

1. Full medical history taking
2. Full clinical examination, APACHE II score on admission
3. Electrolytes panel daily on ICU admission
4. Estimate the duration of stay at ICU Also all selected individuals will be sectioned into groups regarding sites of collection (surgical ICU, CCU and medical ICU). All collected individuals will be sectioned regarding electrolytes imbalance into mild, moderate and severe groups

DETAILED DESCRIPTION:
Study Procedures: All selected individuals will be suffering from electrolyte imbalance (EI) with the following data will be obtained:

o Measurements:

1. Demographic data: age - gender - BMI - electrolytes data on ICU admission
2. Vital data: heart rate - respiratory rate - blood pressure measurement - Oxygen saturation - Urinary output - Temp +/- CVP measurement.
3. Lab.: "CBC - Kidney function tests - liver function tests - ABG - levels of serum sodium, potassium, magnesium, phosphorus, ionized calcium and chloride", with maximum 5 mm blood sampling per day. Serum-sodium levels will be corrected for serum-glucose by lowering the sodium concentration by 2.4 mmol/L for every 100 mg/dl increase in glucose. Corrected Sodium = Measured sodium + 0.016 (Serum glucose - 100) A correction formula was also used to calculate albumin-corrected calcium levels (mmol/L) Corrected Calcium = (0.8 (Normal Albumin - Pt's Albumin)) + Serum Ca
4. APACHE II score
5. Comorbidities
6. Complications: AKI- Acute myocardial infarction
7. Duration of ICU stay
8. Duration of hospital stay
9. Outcome (regarding eventual complications: AKI- Acute myocardial infarction)

ELIGIBILITY:
Inclusion Criteria:

- All patients admitted to medical ICU, surgical ICU and CCU suffering from electrolyte imbalance (EI) over 18 years with the comorbid conditions :

1. Hypertension
2. Heart failure
3. Chronic chest diseases
4. Cancers
5. Chronic kidney disease
6. Diabetes mellitus
7. Cardiac dysrhythmias
8. Pneumonia
9. Sepsis
10. Dehydration
11. Critical bones fractures

Exclusion Criteria:

* Patients with

  1. Age less than 18 year old
  2. Patient or his 1st degree relatives refuse to participate
  3. Patients without electrolytes data
  4. Current smoking

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: critically ill Egyptian patients
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-09-26 (Actual); Primary Completion 2024-08-08 (Estimated); Study Completion 2024-08-08 (Estimated)

PRIMARY OUTCOMES:
impact of electrolytes imbalances for general health status | 1 year
  Laboratory: levels of serum sodium "mmol/L", potassium "mmol/L", magnesium "mg/dl", phosphorus "mg/dl", ionized calcium "mmol/L" and chloride "mmol/L", with maximum 5 mm blood sampling per day. Serum-sodium levels will be corrected for serum-glucose by lowering the sodium concentration by 2.4 mmol/L for every 100 mg/dl increase in glucose.
  Corrected Sodium = Measured sodium + 0.016 (Serum glucose - 100). A correction formula was also used to calculate albumin-corrected calcium levels (mmol/L).
  Corrected Calcium = (0.8 (Normal Albumin - Pt's Albumin)) + Serum Ca

SECONDARY OUTCOMES:
impact of electrolytes imbalances for hospital stay | 1 year
  calculation of hospital admission days and correlations with records of serum electrolytes results per admission

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sadek, MD candidate, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT06097104/Prot_000.pdf
  • Informed Consent Form (2023-09-26): https://cdn.clinicaltrials.gov/large-docs/04/NCT06097104/ICF_001.pdf